CLINICAL TRIAL: NCT06626789
Title: A Multi-center, Patient-blinded and Investigator-blinded, Randomized, Parallel-group, Superiority Study to Compare the Efficacy of Four Sessions of Amygdala fMRI-BOLD Neurofeedback With Yoked Sham-control Neurofeedback in the Treatment of Dysregulated Affect in Borderline Personality Disorder
Brief Title: Brain Signal Training to Enhance Affect Down-regulation
Acronym: BrainSTEADy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: University Medical Center Freiburg (Other); University of Giessen (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BrainSTEADy
Record Dates: First submitted 2024-09-16; First posted 2024-10-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Borderline Personality Disorder
Keywords: Neurofeedback; fMRI; Neuroimaging; Amygdala; Affect instability; Emotion
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Clinical Research Organization (sub-contractor) responsible for interim analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Real-time functional Magnetic Resonance Imaging (fMRI) neurofeedback from the Blood Oxygenation Level Dependent (BOLD) signal of the amygdala
  Interventions: Biological: Amygdala neurofeedback
- Control group (Experimental): Feedback that is less correlated with amygdala BOLD signal
  Interventions: Behavioral: Sham neurofeedback

INTERVENTIONS:
Biological: Amygdala neurofeedback — Real-time fMRI neurofeedback from amygdala's blood oxygenation level dependent (BOLD) signal + negative emotional picture viewing. Instruction to regulate feedback via down-regulation of one's emotional response.
  Arms: Intervention group
Behavioral: Sham neurofeedback — Recorded neurofeedback from a different participant + negative emotional picture viewing. Instruction to regulate feedback via down-regulation of one's emotional response.
  Arms: Control group

SUMMARY:
Individuals with Borderline Personality Disorder (BPD) experience intensive, instable negative emotions. Hyperactivity of the amygdala is assumed to drive exaggerated emotional responses in BPD. Neurofeedback is an endogenous neuromodulation method to address the imbalance of neural circuits. Downregulation of amygdala hyperactivation with neurofeedback may ameliorate dysregulated emotions in BPD. The BrainSTEADy trial is designed to determine whether amygdala-fMRI-BOLD neurofeedback has a specific effect on affect instability in BPD beyond nonspecific benefit.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is characterized by self-mutilation, suicidality, and severe interpersonal disturbances. These symptoms reflect pervasive emotion regulation problems. On the neural level, BPD patients show an inflated amygdala response to emotional cues. In addition, they have reduced neural control of the amygdala. The amygdala controls emotional experience and behavior. Therefore, current psychobiological theories consider amygdala hyper-activity a causal mechanism for emotional overreaction in BPD.

Functional magnetic resonance imaging (fMRI) allows the recording of activation in subcortical brain regions, such as the amygdala, in real time. Live feedback from brain activation (e.g. via a thermometer with the temperature reflecting the degree of activation) allows one to learn the voluntary control of the brain. Dubbed "neurofeedback" (NF), the method can result in long-lasting changes in neural activation patterns. NF allows precise targeting of dysfunctional neuro-circuitries that relate to clinical symptoms.

The project proposed here investigates the clinical effectivity of fMRI-based amygdala-NF training in BPD. In total, 164 patients will participate in four training sessions provided by four study centers: Tuebingen, Freiburg, Giessen, and Mannheim. The training aims to reduce affective instability in everyday life, which is assessed primarily by ambulatory assessment before and after treatment. During NF sessions, patients receive feedback from the BOLD (Blood Oxygenation Level Dependent) signal recorded in the amygdala while they view pictures with negative emotional content. The amygdala responds to these pictures with an activation increase. The patient observes the amygdala responding, illustrated via increased temperature in a thermometer beside the picture. The task is to decrease temperature. The procedure should teach patients to master overreaction at an early stage of neural emotion processing.

To assess the effectivity of amygdala-NF, a control group receives non-veridical feedback from a different patient. The investigators expect a significant reduction in affective instability with amygdala-NF. In addition, the investigators expect a greater reduction in affective instability in the amygdala-NF group versus the control group.

The trial will go through two stages of recruitment. Stage 1 is reached after recruitment of 82 participants. An interim analysis will be conducted. Depending on the results of the interim analysis, the trial will enter stage 2, ie. recruitment of the full number of planned participants.

Results from this study enable assessment of clinical efficacy of amygdala-NF. In the future, NF could serve as a precise tool for person-centered treatment of affective instability symptoms in mental disorders with severe emotion regulation problems such as BPD.

ELIGIBILITY:
Stage 1: 82 patients, stage 2: 82 patients Inclusion Criteria

1. 18-65 years
2. Diagnosis of Borderline Personality Disorder
3. Insufficient response to ≥2 therapies.
4. Sufficient German language skills to give informed consent to the study, to understand questions posed by used instruments, and capable of completing the fMRI tasks
5. Ability of subject to understand character and individual consequences of clinical investigation
6. Written informed consent (must be available before enrollment in the clinical investigation)
7. For women of childbearing potential (WOCBP) adequate contraception.

Exclusion Criteria

1. Treatment with benzodiazepines within 7 days prior the initial screening
2. Current alcohol or substance dependence
3. Meeting the diagnostic criteria for a psychotic disorder or schizophrenia (life-time), as determined by clinical interview at initial screening
4. Current or history of significant neurological condition (such as stroke, traumatic brain injury, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack)
5. Significant visual impairment that might interfere with the performance of the behavioural tasks or fMRI tasks
6. Change of treatment (psychopharmacologic, psychological) 2 weeks prior to or during the study participation
7. Treatment with any neurofeedback three months prior to or during the study participation.
8. Unable or unwilling to comply with study procedures, including study prohibitions and restrictions
9. History of claustrophobia or inability to tolerate scanner environment
10. Fulfilling any of the MRI contraindications on the standard site radiography screening questionnaire (e.g. history of surgery involving metal implants)
11. Clinically relevant structural brain abnormality as determined by prior MRI scan
12. Planned medical treatment within the study period that might interfere with the study procedures
13. Participants deemed to be at significant risk of serious violence or suicide
14. BMI of 16.5 or lower
15. Participation in other clinical trials or observation period of competing trials, respectively
16. Previous participation in this trial
17. Pregnancy and lactation
18. Held in an institution by legal or official order
19. Legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Affect Intensity, change from T0 to T1 | Completion of T0 EMA sampling within 12 days before first NF session. Start of T1 EMA sampling within 1 week after last NF session.
  Mean score of negative affect scale measured via experience sampling using ecological momentary assessment (EMA). Scale can take values from 1 to 7, high values mean higher affect intensity. EMA is conducted across 4 consecutive days, including a full weekend, when patients carry a smartphone that runs the EMA app. The app sends an auditory signal every hour, starting at 9 AM until 9 PM, to remind the patient to fill out the items.

SECONDARY OUTCOMES:
Affect Intensity, change from T0 to T2 | Completion of T0 EMA sampling within 12 days before first NF session. Start of T2 EMA sampling within 14-16 weeks after last NF session.
  Mean score of negative affect scale measured via experience sampling using ecological momentary assessment (EMA). Scale can take values from 1 to 7, high values mean higher affect intensity. EMA is conducted across 4 consecutive days, including a full weekend, when patients carry a smartphone that runs the EMA app. The app sends an auditory signal every hour, starting at 9 AM until 9 PM, to remind the patient to fill out the items.
Borderline Symptom Severity, change from T0 to T1 and T0 to T2 | T0 assessed before first NF session (within 1-3 weeks). T1 assessed after last NF session (within 2-4 weeks). T2 assessed within 14-16 weeks after last NF session.
  Zanarini Rating Scale for BPD, interview version (ZAN-BPD) total score. Total score can take values 0-36 with higher values meaning higher symptom burden.
Amygdala response, change from T0 to T1. | Time Frame: T0 assessed at Baseline. T1 assessed at Post-Assessment immediately after treatment.
  BOLD-fMRI response in the amygdala to negative stimuli in the view-condition, during NF session 1, run 1, vs. last NF session, last run.
Amygdala self-regulation, change from T0 to T1. | Time Frame: T0 assessed at Baseline. T1 assessed at Post-Assessment immediately after treatment.
  BOLD-fMRI response in the amygdala to negative stimuli in the regulate-condition, during NF session 1, run 1, vs. last NF session, last run.
Improvement in quality-adjusted life years (QALY), change from T0 to T3 | T0 assessed before first nf session (within 1-3 weeks). T3 assessed 6 months after last NF session.
  We measure health-related quality of life with the AQoL-6D (Centre for Health Economics, Monash University, 2016), a multi attribute utility instrument frequently used in health economic evaluations. We elicit quality adjusted life years (QALYs) from the AQoL-6D unweighted scorings by using established value sets. The derived QALYs range from 0.00 to 1.00, where 0.00 represents death and 1.00 a year in perfect health. We combine effects (QALYs) and costs of utilization between groups to receive incremental cost-effectiveness ratios (ICER). Thus, we are able to present costs per QALY for the neurofeedback intervention to inform stakeholders in health care about reimbursement decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Paret-Voigt, Dr., Principal Investigator — ZI Mannheim
Locations (6):
- Germany (6):
  - University clinic Freiburg, Freiburg im Breisgau
  - University clinic Giessen, Giessen
  - University Clinic Halle (Saale), Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Central Institute of Mental Health, Mannheim
  - University Clinic Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized and de-identified data will be uploaded to a data repository hosted by University of Heidelberg (heiDATA).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available within 1 year after completion of data collection. Data will be available for at least 10 years.
Access Criteria: IPD can be shared with researchers who are located in countries with a data protection level that is equivalent with the EU-GDPR. Researcher have to request access at the repository website.

REFERENCES:
- [Background] Zaehringer J, Ende G, Santangelo P, Kleindienst N, Ruf M, Bertsch K, Bohus M, Schmahl C, Paret C. Improved emotion regulation after neurofeedback: A single-arm trial in patients with borderline personality disorder. Neuroimage Clin. 2019;24:102032. doi: 10.1016/j.nicl.2019.102032. Epub 2019 Oct 16. PMID 31795041
- [Background] Paret C, Kluetsch R, Zaehringer J, Ruf M, Demirakca T, Bohus M, Ende G, Schmahl C. Alterations of amygdala-prefrontal connectivity with real-time fMRI neurofeedback in BPD patients. Soc Cogn Affect Neurosci. 2016 Jun;11(6):952-60. doi: 10.1093/scan/nsw016. Epub 2016 Feb 1. PMID 26833918
- [Background] Paret C, Kluetsch R, Ruf M, Demirakca T, Hoesterey S, Ende G, Schmahl C. Down-regulation of amygdala activation with real-time fMRI neurofeedback in a healthy female sample. Front Behav Neurosci. 2014 Sep 18;8:299. doi: 10.3389/fnbeh.2014.00299. eCollection 2014. PMID 25278851
- [Derived] Paret C, Jindrova M, Kleindienst N, Eck J, Breman H, Luhrs M, Barth B, Ethofer T, Fallgatter AJ, Goebel R, Hoell A, Lockhofen D, Reinhold AS, Maier S, Matthies S, Mulert C, Schonholz C, van Elst LT, Schmahl C. A randomised controlled trial of amygdala fMRI-neurofeedback versus sham-feedback in borderline-personality disorder - systematic literature review and introduction to the BrainSTEADy trial. BMC Psychiatry. 2025 Jul 8;25(1):687. doi: 10.1186/s12888-025-07000-1. PMID 40629288
- See also: Trial recruitment website — https://www.borderline-neurofeedback.de/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT06626789/Prot_SAP_003.pdf